CLINICAL TRIAL: NCT06541548
Title: Comparison of Bone Microarchitecture Analysed by High Resolution Peripheral Microscanner (HR-pQCT) and Peripheral Microscanner (pQCT) in Pathologies With Bone Loss and/or Muscle Loss
Brief Title: Comparison of Bone Microarchitecture Analysed by HRpQCT and pQCT in Pathologies With Bone Loss and/or Muscle Loss
Acronym: MICROS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24CH080; ANSM (Other: 2024-A01130-47)
Record Dates: First submitted 2024-07-25; First posted 2024-08-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis Risk; Bone Loss
Keywords: Bone microarchitecture; Bone fragility; osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Describe bone quality and quantity with HR-pQCT, pQCT and DEXA in the group of patients at risk of osteoporosis.
  Interventions: Device: HR-pQCT; Device: pQCT; Device: DEXA
- Control group (Experimental): Describe the quality and quantity of bones with HR-pQCT, pQCT and DEXA in the group of patients not at risk of osteoporosis.
  Interventions: Device: HR-pQCT; Device: pQCT; Device: DEXA

INTERVENTIONS:
Device: HR-pQCT — Xtreme CT® device is a high resolution peripheral quantitative computed tomography (HR-pQCT) used to measure bone density and quantify the bone architecture to 3D at the extremities of the human body.
  For the study, the device will be used to assess bone density and microarchitecture at the forearm and shin for a systemic effect. In rheumatoid arthritis, bone density and microarchitecture will also be measured at the metacarpophalangeal.
Device: pQCT — Peripheral Quantitative Computed Tomography (pQCT) will be performed and measure bone and muscle parameters.
Device: DEXA — The Lunar Dual Energy X-ray Absorptiometry (DEXA) is a third generation multi-captor DEXA device that allow short duration measurements. It measures Bone Mineral Density (BMD) at the spine and the femoral neck.

SUMMARY:
The study aims to utilize medical devices, such as the Xtreme CT and XCT 3000, to assess bone and muscle microarchitecture for various pathologies. The devices provide crucial data on bone and muscle density, aiding in understanding fracture risks associated with conditions like rheumatoid arthritis and neurological disorders. Current methods like DXA scanning have limitations in predicting fracture risks accurately due to their inability to assess cortical and trabecular microstructure. The study emphasizes the importance of evaluating cortical porosity and trabecular volume loss, especially in conditions like post-menopausal osteoporosis and sarcopenia. Additionally, it explores the impact of neurological disorders, renal insufficiency, and endocrinopathies on bone health. Furthermore, the study aims to establish a control group to differentiate pathological changes from age-related variations. Expected outcomes include a comprehensive understanding of bone microarchitecture alterations across various pathologies and the potential to improve fracture risk estimation beyond conventional methods like DEXA scanning. Ultimately, the study anticipates facilitating better management strategies to reduce fracture risks associated with these conditions.

ELIGIBILITY:
Inclusion Criteria:

For the patients:

Women or men treated at the Saint-Etienne University Hospital and presenting an osteoporotic risk with one of the following associated pathologies:

* Osteoporosis defined by: History of a documented brittle bone fracture
* Bone fragility: Patient with indication for bone densitometry but no history of fracture
* Inflammatory joint disease:

  * Rheumatoid arthritis
  * Spondyloarthritis
* Chronic kidney disease
* Endocrinopathies:

  * Primary hyperparathyroidism
  * Constitutional thinness
  * Anorexia nervosa
  * Obesity (BMI >30)
  * Sarcopenia
* Neuropathies - Parkinson's disease

For the controls:

Acute episode of spinal or radiculalgia (less than one month old) with corticosteroid treatment of less than 1 month Signature of written consent

Exclusion Criteria:

* No sign written consent

For the controls:

* Medications inducing bone loss:
* anti-aromasin or GnRH agonist for at least 6 months,
* corticosteroids (dose ≥ 5 mg/d for 6 months)
* anti-epileptic drugs: carbamazepine, phenobarbital, phenytoin, primidone, valproic acid for at least 6 months)
* History of fracture due to bone fragility
* Taking bone-targeting medication (biphosphonate, teriparatide, strontium ranelate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2035-05 (Estimated); Study Completion 2035-05 (Estimated)

PRIMARY OUTCOMES:
total volumetric mineral density by HR-pQCT | Day 1
  Describe total volumetric mineral density (mg/ccm HA) as a function of pathologies
trabecular volumetric mineral density by HR-pQCT | Day 1
  Describe trabecular volumetric mineral density (mg/ccm HA) as a function of pathologies.
Cortical volumetric mineral density by HR-pQCT | Day 1
  Describe cortical volumetric mineral density (mg/ccm HA) as a function of pathologies.
Describe number of trabeculae by HR-pQCT | Day 1
  Number of trabeculae (1/mm) as a function of pathologies.
Trabecular thickness by HR-pQCT | Day 1
  Describe trabecular thickness (mm) as a function of pathologies.
cortical thickness (mm) by HR-pQCT | Day 1
  Describe cortical thickness (mm) as a function of pathologies.
trabecular separation by HR-pQCT | Day 1
  Describe trabecular separation (mm) as a function of pathologies.
cortical porosity by HR-pQCT | Day 1
  Describe cortical porosity (%) as a function of pathologies.

SECONDARY OUTCOMES:
Total bone mineral content with pQCT | Day 1
  Total bone mineral content (mg)
Total bone surface with pQCT | Day 1
  Total bone surface (mm2)
Total bone density with pQCT | Day 1
  Total bone density (mg/mm3)
Cortical and trabecular density with pQCT | Day 1
  Cortical and trabecular density (mg/mm3)
bone resistance index with pQCT | Day 1
  bone resistance index (g2/mm)
Bone density by DEXA | Day 1
  Parameter measured by DEXA is Bone Mineral Density (BMD, g/cm2).
volumetric mineral density with HR-PQCT | Day 1
  Total volumetric mineral density (mg/ccm HA)
Trabecular volumetric mineral density with HR-PQCT | Day 1
  Trabecular volumetric mineral density (mg/ccm HA)
Cortical volumetric mineral density with HR-PQCT | Day 1
  Cortical volumetric mineral density (mg/ccm HA).

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No